CLINICAL TRIAL: NCT00189462
Title: A Pilot Study to Evaluate the Efficacy of Montelukast in the Treatment of Acute Otitis Media (AOM) in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deborah Gentile (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Deborah Gentile, Co- Investigator, Asthma & Allergy Dept, West Penn Allegheny Health System
Organization: West Penn Allegheny Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC - 3643
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Acute Otitis Media; Otitis Media; Ear Infection
Keywords: Ear Infections; Otitis Media
MeSH Terms: conditions — Otitis Media; Otitis | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): Treatment with montelukast for 4 months (4 mg per day)
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Treatment with placebo for 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast
  Arms: Montelukast
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this pilot study is to evaluate the efficacy of treatment with montelukast as compared to placebo in the prevention of recurrence of acute Otitis media (AOM)

DETAILED DESCRIPTION:
Otitis media (OM) is one of the most common childhood disorders requiring physician care and has been associated with an alarming rise in prevalence. Certain children are prone to recurrent episodes of acute Otitis media (RAOM) and/or the development of chronic Otitis media with effusion (COME). Because medical therapy with antibiotics, antihistamines, decongestants and corticosteroids has no demonstrable efficacy, the mainstay of treatment is surgical intervention, which is quite expensive and exposes patients to risks of general anesthesia. The objective of this pilot study is to evaluate the efficacy of treatment with montelukast as compared to placebo in the prevention of recurrence of acute Otitis media (AOM)

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 months to 5 years old.
* Diagnosis of current AOM

Exclusion Criteria:

* Presence of primary or secondary immunodeficiency, craniofacial abnormality, cleft palate, anatomic predisposition, major congenital anomaly or syndrome, or severe systemic disease
* Use of:

  * Any investigational medications within the past 30 days, systemic or oral or nasal steroids within the past 30 days
  * Accolate® in the past 7 days
  * Antibiotics within the past week, except for Zithromax®, which will be 21 days
  * Long acting second generation antihistamines (i.e., Claritin®, Clarinex®, Allegra® and Zyrtec®) within the past 72 hours.
* No known allergy to either montelukast or amoxicillin/clavulanate
* Have not responded to Augmentin® in the past

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2004-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoner, MD, Principal Investigator — West Penn Allegheny Health System
Locations (2):
- United States (2):
  - Bellevue Pediatric Associates, Bellevue, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast: Treatment with montelukast for 4 months (4 mg per day)
  Montelukast
Period: Overall Study
Arm/Group | Montelukast | Placebo
Started | 50 | 49
Completed | 27 | 28
Not Completed | 23 | 21
Not completed — Lack of Efficacy | 5 | 1
Not completed — Lost to Follow-up | 18 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Placebo | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 49 | 99
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 26 | 29 | 55
Region of Enrollment [Number; unit: participants] — All subjects were enrolled in the Pittsburgh area
  participants
    United States | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Otitis Media
Time Frame: 16 weeks
Measure: Number; unit: participants with AOM
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 50 | 49
participants with AOM | 30 | 27

ADVERSE EVENTS:
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 16/50 | 15/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast (N=50) | Placebo (N=49)
Diarrhea (General disorders) | 5 | 6
Vomiting (General disorders) | 3 | 2
Rash (General disorders) | 0 | 3
Cold/Upper Respiratory Infection (General disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No